CLINICAL TRIAL: NCT07351110
Title: Improving Cervical Cancer Prevention Among Women Living With Chronic Conditions. Aim 3: Assess the Feasibility and Acceptability of the PINPOINT Intervention.
Brief Title: Improving Cervical Cancer Prevention Among Women Living With Chronic Conditions.
Acronym: PINPOINT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IRB202500780; 1K01CA292583-01 (NIH)
Record Dates: First submitted 2026-01-16; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Diabetes; Cervical Cancer (Early Detection); Obesity & Overweight
Keywords: cervical cancer screening; self-collection; self-sampling
MeSH Terms: conditions — Diabetes Mellitus; Uterine Cervical Neoplasms; Obesity; Overweight | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): PINPOINT intervention arm will entail assigning patients to a patient navigator to assist them with screening reminders and address any barriers they have to screening, education on cervical cancer screening, and patients will also be offered the opportunity to self-collect their sample for cervical cancer screening.
  Interventions: Behavioral: patient navigation and self-collection
- Control Arm (No Intervention): No intervention arm, patients will receive reminders for screening according to current clinical practice

INTERVENTIONS:
Behavioral: patient navigation and self-collection — Patients will receive a combination of patient navigation, education, and cervical cancer self-collection sampling as part of the intervention to support cervical cancer screening.
  Other Names: self-collection; self-sampling; patient navigation
  Arms: Intervention

SUMMARY:
Our overarching goal is to adapt and test the PINPOINT intervention -PatIent Navigation for the Prevention of CervIcal CaNcer inTervention. We will test the PINPOINT intervention among patients with high-risk profiles for cervical cancer who do not meet the recommended screening for cervical cancer.

DETAILED DESCRIPTION:
We will test the PINPOINT intervention among patients with high-risk profiles for cervical cancer who do not meet the recommended screening for cervical cancer. We will use the six steps of the Intervention Mapping approach to guide the process of testing the intervention. This project aligns with the current efforts at the University of Florida Health Cancer Institute (UFHCI) and UF Health Internal Medicine to improve cervical cancer screening rates among under-screened women. We will partner with these efforts to test the PINPOINT intervention. Project CONTINUITY (Connecting You to Care in the Community) at UFHCI, Office of Community Outreach and Engagement (COE), is working to increase adherence to cervical screening and follow-up by; (1) providing personalized approaches to improve adherence through the combined use of patient choice for the initial screening method, community clinical navigators (CCN) and community health workers (CHWs), customized messages and support for patient portal access for test results, and (2) implementing strategies to address non-medical drivers that may influence an individual's ability to adhere to the screening, with an initial focus on removing transportation barriers through the use of a mobile outreach clinic (MOC).

Currently, a patient navigator supervised by Dr. Dianne Goede identifies patients who have an upcoming office visit and are due for cervical cancer screening at UF Health Internal Medicine. The patient navigator outreaches the patient, reminds them of their overdue status for cervical cancer screening and the importance of cervical cancer screening, and inquires if they are agreeable to complete screening at the scheduled office visit. We will reach out to patients who remain unscreened for cervical cancer 2 months after their scheduled visit with UF Health Internal Medicine. We will obtain a list of patients from the UF Health Consent2Share database. Patients who agree to participate in our study will be randomized to either receive the PINPOINT intervention (self-collection test with patient navigation) or standard of care (reminder to screen from UF Health Internal Medicine). We will use the sealed envelope randomization method to assign participants to either treatment or control groups right after intake.

We will pilot the PINPOINT intervention at UF Internal Medicine clinics and use Proctor's Framework for Implementation Outcomes to evaluate the intervention. Changes will be made to the intervention protocol and tested in a future randomized trial with a larger sample. Hypothesis: PINPOINT will meet the needs of women living with socioeconomic challenges, T2D, and obesity, and will align with the clinical workflow. PINPOINT will be appropriate, feasible and acceptable.27 Outcome: The PINPOINT intervention will have positive outcomes in terms of feasibility and acceptability among patients.

ELIGIBILITY:
Inclusion Criteria:

The following eligibility criteria will be used to determine inclusion into the study:

1. Using the American Cancer Society (ACS) screening recommendations, adults aged over the age of 25 will be eligible
2. Active UF Internal Medicine patient and has had an appointment in the last 2 months.
3. Assigned sex at birth is female
4. Have Obesity or Type 2 Diabetes
5. Not currently pregnant (self-report)
6. Have not given birth in the prior 12 weeks
7. No previous history of cervical cancer
8. No previous history of a hysterectomy
9. Have not undergone cancer screening in the past 3 years or more
10. Reside in the UFHCI Catchment Area (Alachua, Baker, Bradford, Citrus, Clay, Columbia, Dixie, Gadsden, Gilchrist, Hamilton, Jefferson, Lafayette, Lake, Leon, Levy, Madison, Marion, Putnam, Sumter, Suwannee, Taylor, UnioF1n, or Wakulla County).
11. Have a mobile phone or access to a mobile phone that can be used to receive messages, or a valid email address.
12. Are not currently scheduled to receive cervical cancer screening via clinician sampling (pap smear).

Exclusion Criteria:

* Previous history of cervical cancer
* Total hysterectomy
* Pregnant

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-12-24 (Estimated)

PRIMARY OUTCOMES:
Cervical cancer screening | within 6 months
  receiving cervical cancer screening either via self-collection, pap smear, or hpv testing

SECONDARY OUTCOMES:
Acceptability | from enrollment until they complete screening or at the end of the trial at 6 months
  How agreeable or satisfactory participants find the intervention or implementation strategy. Questions include, HPV Self-Collection meets my approval, HPV Self-Collection is appealing to me, I like HPV Self-Collection, and I welcome HPV Self-Collection. Participants will fill a 4 point likert scale for each, (completely disagree, disagree, neither agree not disagree, agree, completely agree).
Appropriateness | from enrollment until they complete screening or at the end of the trial at 6 months
  The perceived fit or compatibility of the intervention for a specific setting, provider, or consumer, or to address a problem. Questions include, HPV Self-Collection seems fitting, HPV Self-Collection seems suitable, HPV Self-Collection seems applicable., and HPV Self-Collection seems like a good match. Participants will fill a 4 point likert scale for each, (completely disagree, disagree, neither agree not disagree, agree, completely agree).
Feasibility measure | from enrollment until they complete screening or at the end of the trial at 6 months
  - The extent to which an intervention can be successfully used in a given setting. Questions include, HPV Self-Collection seems implementable, HPV Self-Collection seems possible, HPV Self-Collection seems doable, and HPV Self-Collection seems easy to use. Participants will fill a 4 point likert scale for each, (completely disagree, disagree, neither agree not disagree, agree, completely agree).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UF Health Internal Medicine, Gainesville, Florida
  - University of Florida, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Deidentified data will be available after the results of the study are published.

REFERENCES:
- [Background] Mkuu RS, Staras SA, Szurek SM, D'Ingeo D, Gerend MA, Goede DL, Shenkman EA. Clinicians' perceptions of barriers to cervical cancer screening for women living with behavioral health conditions: a focus group study. BMC Cancer. 2022 Mar 9;22(1):252. doi: 10.1186/s12885-022-09350-5. PMID 35264120
- [Background] Mkuu RS, Tohme S, Rivero-Mendoza D, Salloum RG, Goede D, Bruggeman B, Nicholson K, Hall JM, Bylund C, Woodard JN, Hensley J, Shenkman EA, Donahoo WT, Mulugeta A, Hernandez M, Staras SA. Improving Patient Education Materials for HPV Self-Collection: Insights from Women at High Risk of Developing Cervical Cancer. Cancer Manag Res. 2025 Dec 24;17:3273-3284. doi: 10.2147/CMAR.S552282. eCollection 2025. PMID 41467104
- [Background] Mkuu RS, Staras SA, Chakrabarti C, Hall J, Harvey I, Salloum RG, Barrow S, Ortega S, Woodard J, Seals K, Rawls A, Meduri Y, Donahoo WT, Goede DL, Shenkman EA. Acceptability of HPV self-collection: A qualitative study of Black women living with type II diabetes and social vulnerability. J Clin Transl Endocrinol. 2024 Feb 25;35:100331. doi: 10.1016/j.jcte.2024.100331. eCollection 2024 Mar. PMID 38444842
- See also: Study Funding Information — https://reporter.nih.gov/search/TYyuoez0OUWufZdq8tAD-A/project-details/10949284